CLINICAL TRIAL: NCT02609841
Title: POtassium and Cardiac Rhythm Trends in MaintENance HemoDialysis (PORTEND): A Multicenter, Prospective, Observational Study
Brief Title: POtassium and Cardiac Rhythm Trends in MaintENance HemoDialysis: A Multicenter, Prospective, Observational Study
Acronym: PORTEND
Status: Completed | Type: Observational
Sponsor: ZS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ZS-008
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Cardiac rhythm remote monitoring system: Subjects use non-invasive wearable BodyGuardian remote monitoring system throughout 12 days of study.
  Interventions: Device: Cardiac rhythm remote monitoring system

INTERVENTIONS:
Device: Cardiac rhythm remote monitoring system — Non-invasive wearable remote cardiac rhythm monitoring system used throughout 12 days of study.
  Other Names: BodyGuardian

SUMMARY:
This study assesses serum potassium and cardiac rhythm trends in subjects with end stage renal disease (ESRD) who are on 3 times weekly maintenance hemodialysis for at least 60 days. Dialysate K (relative potassium concentration in dialysate) must be stable for 2 weeks prior to enrollment.The number of subjects on 3K or higher dialysate will be limited to 60, with the remainder of the subjects on 1K or 2K dialysate.

DETAILED DESCRIPTION:
This study assesses serum potassium and cardiac rhythm trends in subjects with end stage renal disease (ESRD) who are on 3 times weekly maintenance hemodialysis for at least 60 days. Approximately 240 Subjects who meet the eligibility criteria and sign the informed consent form can be enrolled in the study, after which a subject number will be assigned. The number of subjects on 3K or higher dialysate will be limited to 60, with the remainder of the subjects on 1K or 2K dialysate. Baseline data will be collected including subject demographics, dialysis prescription, and symptom assessment. In addition, results of clinical laboratory tests and urea reduction ratio (URR), dialyzer clearance-time-volume of distribution of urea (Kt/V), and intact parathyroid hormone (PTH) obtained within the 4 weeks prior to the first dialysis treatment on Study Day 1 will be collected from regular monthly labs to establish baseline.

Subjects will be assessed in the dialysis clinic/research center over a period of 12 days. Subjects will start the study on the first day of a given week's dialysis regimen (ie, Monday or Tuesday). Subjects who are on a Monday, Wednesday, and Friday dialysis schedule will skip the Saturday visit, and subjects who are on a Tuesday, Thursday, and Saturday dialysis schedule will skip the Sunday visit during the 12-day study duration.

Subjects will undergo blood collection at each visit, including 6 dialysis days and 5 inter-dialysis days. On dialysis days, blood samples will be collected immediately before and at the end of dialysis treatment. During the dialysis treatments on Study Days 1 and 3 only, additional blood samples will be obtained at 30 minutes and 1 hour (± 15 minutes) after the start of dialysis for chemistry. On inter-dialysis days, the dialysis clinic/research center will make an effort to collect blood samples at the same approximate time that dialysis treatment would have started on days of dialysis. Otherwise, samples may be collected when the subject is able to visit the dialysis clinic/research center.

Vital signs including heart rate and blood pressure, and body weight will be collected at each visit. On dialysis days, both pre- and post-dialysis weights will be collected, along with vital signs obtained during dialysis. A specifically designed symptom assessment will also be performed at specified times throughout the study.

The subjects will also undergo cardiac rhythm monitoring using a non-invasive, Food and Drug Administration cleared, wearable device (BodyGuardian® remote monitoring system) throughout the 12 days of participation in the study. This will be used to assess for cardiac arrhythmias, as well as to correlate S-K levels with signal-averaged, processed ECG.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* 18 years of age or older.
* Subject has ESRD and has been stable and compliant (as determined by the investigator) on 3 times weekly maintenance hemodialysis for at least 60 days; the number of subjects on 3K or higher dialysate will be limited to 60, with the remainder of the subjects on 1K or 2K dialysate. Dialysate K must be stable for 2 weeks prior to enrollment.
* Hemoglobin > 9 g/dL.
* Able to undergo peripheral venous sticks for blood draws on inter-dialysis days, or the dialysis/research team is able to use the dialysis access for blood draws on those days.
* Subject or subject's caregiver at home can read and understand English and has the ability to use the BodyGuardian remote monitoring system.

Exclusion Criteria:

* Pregnancy. Sexually active women of child-bearing potential must have a negative pregnancy test before starting the study on Study Day 1. Women who are surgically sterile or those who are postmenopausal for at least 2 years are not considered to be a childbearing potential.
* Subjects or bed partners with implanted pacemakers or defibrillators.
* Known skin allergies or sensitivities to acrylic, hydrogel or silicone adhesives.
* Fragile skin.
* Participation in another clinical trial which may impact the results of this study.
* Subjects who, in the opinion of investigator, are unable to perform the tasks associated with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects has ESRD and has been stable and compliant (as determined by the investigator) on 3 times weekly maintenance hemodialysis for at least 60 days.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Chair — ZS Pharma, Inc.
Locations (9):
- United States (9):
  - Los Angeles, California
  - San Jose, California
  - Denver, Colorado
  - Evergreen Park, Illinois
  - Rochester, Minnesota
  - Flushing, New York
  - Chattanooga, Tennessee
  - Lufkin, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with end stage renal disease on maintenance hemodialysis took part in the study at 17 sites in the United States.
Pre-assignment Details: Cardiac rhythm was monitored using a 24-hour non-invasive, wearable device (BodyGuardian® remote monitoring system) throughout the study to assess for cardiac arrhythmias was to be worn by patients. One site did not perform cardiac rhythm monitoring.
Groups:
- Enrolled Study Population: All patients who were enrolled in the study
Period: Overall Study
Arm/Group | Enrolled Study Population
Started | 240
Completed | 212
Not Completed | 28

BASELINE CHARACTERISTICS:
Population: Baseline data was summarized only for those patients who received all 6 hemodialysis (HD) treatments over 12 days; 28 patients did not complete all treatments and are excluded from baseline population.
Groups:
- <3 K Dialysate Patients: Patients on <3 K dialysate and received all 6 hemodialysis treatments over 12 days.
- ≥3K Dialysate Patients: Patients on ≥3K dialysate who received all 6 hemodialysis treatments over 12 days
- Total: Total of all reporting groups
Arm/Group | <3 K Dialysate Patients | ≥3K Dialysate Patients | Total
Number analyzed (Participants) | 179 | 33 | 212
Age, Customized [Mean (Standard Deviation); unit: Years] | 56.9 (12.4) | 58.5 (12.4) | 57.1 (12.5)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 64 | 13 | 77
  Male | 115 | 20 | 135

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pre-dialysis HK After the LIDP in <3K Dialysate Patients
Description: Incidence of pre-dialysis hyperkalemia (HK) in patients after the long inter-dialytic period (LIDP) in patients on <3K dialysate. Hyperkalemia defined as serum potassium (S-K) >5.0 mEq/L.
Time Frame: 12 Days
Population: Per Protocol Population: all enrolled subjects who receive 6 dialysis treatments within the 12-day study period
Measure: Number; unit: Percent of participants
Groups:
- <3 K Dialysate Patients: Subjects on <3 K dialysate and received all 6 hemodialysis treatments over 12 days.
Arm/Group | <3 K Dialysate Patients
Number analyzed (Participants) | 179
Percent of participants
  Any pre-dialysis HK after LIDP, % | 50
  Pre-dialysis HK after LIDP ( based on mean S-K), % | 37

2. Secondary Outcome: Incidence of Pre-dialysis Hyperkalemia (HK) After the Long Inter-dialytic Period (LIDP) in Patients on ≥3K Dialysate.
Description: Incidence of pre-dialysis hyperkalemia (HK) in patients after the long inter-dialytic period (LIDP) in patients on ≥3K dialysate. Hyperkalemia defined as serum potassium (S-K) >5.0 mEq/L.
Time Frame: 12 days
Population: Per protocol population
Measure: Number; unit: % of patients
Groups:
- ≥3 K Dialysate Patients: Subjects on ≥3 K dialysate and received all 6 hemodialysis treatments over 12 days.
Arm/Group | ≥3 K Dialysate Patients
Number analyzed (Participants) | 33
% of patients
  Any pre-dialysis HK after LIDP, % | 36
  Pre-dialysis HK after LIDP ( based on mean S-K), % | 21

3. Secondary Outcome: Incidence of Cardiac Arrhythmias
Description: Incidence of serious cardiac arrhythmias in patients during the observational period. Serious arrhythmias defined as ventricular tachycardia or > 5 sec pause.
Time Frame: 12 days
Population: Patients who received all 6 hemodialysis treatments and wore Body Guardian Device, a non-invasive wearable remote cardiac rhythm monitoring system
Measure: Number; unit: % of patients
Groups:
- Completed the Study and Wore the Body Guardian: All subjects (<3 K dialysate or dialysate combined) who received all 6 hemodialysis treatments over 12 days and wore the Body Guardian device
Arm/Group | Completed the Study and Wore the Body Guardian
Number analyzed (Participants) | 191
% of patients
  Atrial fibrillation | 51
  Serious arrhythmias | 16

ADVERSE EVENTS:
Description: Due to the observational nature of the study individual adverse events were not collected.
Groups:
- Cardiac Rhythm Monitoring System: Subjects use non-invasive wearable BodyGuardian remote monitoring system throughout 12 days of study.
Arm/Group | Cardiac Rhythm Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZS Pharma has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication